CLINICAL TRIAL: NCT02928887
Title: Light Therapy in Cardiopulmonary Bypass Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Cardiac surgeon collaborator has left the institution
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Matthew Rosengart, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRO16090192
Record Dates: First submitted 2016-10-05; First posted 2016-10-10 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Acute Kidney Injury; Inflammation
MeSH Terms: conditions — Acute Kidney Injury; Inflammation | interventions — Blue Light

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blue light (Experimental): Exposure to high illuminance (1000 lux), blue spectrum (480nm) light for the 24 hour photoperiod prior to surgery and for the 24 hour photoperiod immediately after surgery
  Interventions: Other: Blue light
- Ambient light (No Intervention): Exposure to ambient, white fluorescent light

INTERVENTIONS:
Other: Blue light — Exposure to high illuminance (1000 lux), blue spectrum (480 nm) light for a 24-hour photoperiod immediately before surgery and a 24-hour photoperiod immediately after surgery
  Arms: Blue light

SUMMARY:
The goal of this study is to determine whether or not exposure to blue spectrum light reduces acute kidney injury and systemic inflammation in subjects undergoing cardiopulmonary bypass. Subjects scheduled to undergo cardiopulmonary bypass surgery will be exposed to either bright (1000 lux) blue spectrum (480nm) light or to ambient, white fluorescent light for a 24 hour photoperiod the day prior to surgery and for a 24 hour photoperiod in the immediate postoperative period.

DETAILED DESCRIPTION:
Light modifies the biology and physiology of mammals, including humans. The cellular biology of both the immune system, as well as, the cells comprising tissues and organs (e.g., kidney, liver) are under the regulation of light and exhibit circadian rhythms. Studies show that the severity of organ injury varies with the time of the day, the duration of the day, and the season. This variation is due to the biology of circadian rhythms, and light is the principle environmental cue entraining circadian biology. More recent data suggest that modulating the spectrum of light to which an organism is exposed may therapeutically modulate the cellular response to stress or injury. Specifically, exposure to a short (24 hour) photoperiod of high illuminance, blue spectrum light attenuated liver and kidney injury when animals were subjected to ischemia/reperfusion (I/R), a model in which the blood flow to an organ is temporarily reduced and then restored. A predominant cause of organ injury in this model is the misdirected and exacerbated inflammation of a type of immune cell called the neutrophil. However, blue light inhibited neutrophil infiltration into the ischemic kidney and liver, and thereby reduced inflammation and neutrophil-mediated organ injury.

Cardiopulmonary bypass (CPB) surgery is an operation characterized by excessive inflammation and a high risk of organ injury, particularly acute kidney injury (AKI). Thus, we hypothesize that exposure to blue light, by comparison to standard environmental, white fluorescent light, will reduce inflammation, organ injury and improve the outcome of patients undergoing CPB.

ELIGIBILITY:
Inclusion Criteria:

* age greater than or equal to 18 years
* undergoing cardiopulmonary bypass surgery

Exclusion Criteria:

* Blindness
* Immunocompromised or immunosuppressed state
* Anticipated survival < 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in creatinine concentration | Change in serum creatinine concentration at 24 hours after surgery compared to preoperative baseline creatinine concentration
  The change in serum creatinine after intervention compared to baseline.
Change in blood urea nitrogen (BUN) concentration | Change in serum BUN concentration at 24 hours after surgery compared to preoperative baseline BUN concentration
  The change in serum BUN after intervention compared to baseline.

SECONDARY OUTCOMES:
Inflammation | Change in serum cytokine concentrations comparing serum concentrations at 24 hours after surgery to serum concentrations immediately (with 1 hour) after surgery
  The change in serum concentration of inflammatory mediators after intervention compared to baseline.
all cause mortality | within 28 days after surgery
  Death 28 days after surgery and intervention
duration of ICU stay | within 28 days after surgery
  ICU length of stay 28 days after surgery and intervention
duration of hospital stay | within 28 days after surgery
  Hospital length of stay 28 days after surgery and intervention
Ventilator-free days | within 28 days after surgery
  Cumulative days without mechanical ventilation 28 days after surgery and intervention
Duration of renal replacement therapy | within 28 days after surgery
  Days of dialysis within the first 28 days after surgery and intervention

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Rosengart, MD MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- Presbyterian Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yuan D, Collage RD, Huang H, Zhang X, Kautza BC, Lewis AJ, Zuckerbraun BS, Tsung A, Angus DC, Rosengart MR. Blue light reduces organ injury from ischemia and reperfusion. Proc Natl Acad Sci U S A. 2016 May 10;113(19):5239-44. doi: 10.1073/pnas.1515296113. Epub 2016 Apr 25. PMID 27114521
- [Background] Castro RA, Angus DC, Hong SY, Lee C, Weissfeld LA, Clermont G, Rosengart MR. Light and the outcome of the critically ill: an observational cohort study. Crit Care. 2012 Jul 24;16(4):R132. doi: 10.1186/cc11437. PMID 22827924